CLINICAL TRIAL: NCT02459145
Title: Assessing the Effects of a Clinical Exercise Protocol on Children With Post-concussion Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left Insitution - study no RCT
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS0001
Record Dates: First submitted 2015-05-19; First posted 2015-06-01 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Post Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Graduated Exercise Protocol (Active Comparator): Intervention involves exercise starting at 50% of maximum age-adjusted heart rate (MHR) for 10 minutes (warm-up and Recovery)_ plus 5 minutes of target heart rate per day 5 days a week for 2 weeks, supervised by the athletic trainer or parent. The protocol increases the intensity of target heart rate by 10% MHR and duration of 50% MHR by 2 minutes every 2 weeks if there is no symptom exacerbation. The exercise protocol includes treadmill speed and track minutes per lap conversion, rate of perceived exertion and talk test for each stage of exercise plus total time to execute for 5 days each week.
  Interventions: Behavioral: Graduated exercise protocol
- Rest followed by Protocol (Other): No activity in weeks 1 - 8. In week 9 we will begin their intervention phase as described in graduated exercise protocol
  Interventions: Behavioral: Graduated exercise protocol

INTERVENTIONS:
Behavioral: Graduated exercise protocol — Intervention involves exercise protocols starting at 50% of maximum age-adjusted heart rate (MHR) for 10 minutes (warm-up and Recovery)_ plus 5 minutes of target heart rate per day 5 days a week for 2 weeks, supervised by the athletic trainer or parent. The protocol increases the intensity of target heart rate by 10% MHR and duration of 50% MHR by 2 minutes every 2 weeks if there is no symptom exacerbation.

SUMMARY:
The general consensus in sports medicine demonstrates a graduated return to activity protocol for individuals with post-concussion syndrome. This is commonly practiced but there is insufficient literature to indicate evidence-based practice. This study will provide evidence of the effectiveness of the clinical gradual return to exercise protocols beginning after diagnosis of post-concussion syndrome through standardization and measurement of outcomes.

DETAILED DESCRIPTION:
Concussion is referred to as a mild form of traumatic brain injury (mTBI) that can result in temporary loss of consciousness, memory, or awareness. mTBI can also cause physiologic symptoms such as nausea or vomiting, headaches, vestibulo-ocular dysfunction, and balance errors. The majority of individuals with mTBI will fully recover within a 7-10 day period, although adolescents may require more time to recover than adults. The American Medical Society for Sports Medicine (AMSSM) position statement on concussion management indicates that there are no standardized guidelines for return to school and return to play recommendations involve a graduated activity program once all symptoms have resolved.[1] Treatment varies amongst physicians, but it is widely held that a minimum of 5 days strict rest at home (specifically, no school, work, or physical activity) followed by a stepwise return to activity. Recent articles, however have questioned the validity of strict rest for that many days as for other similar injuries (whiplash) recommendations involve attempts to gradually resume normal activities of daily living.[2]

Individuals whose concussion symptoms do not resolve within 7-10 days are considered to have post concussion syndrome (PCS) which is ill-defined and poorly understood, however the AMSSM describes the benefit of supervised progressive exercise programs that increase tolerance as symptoms permit. The protocols in the literature for adults involve assessing the maximum threshold at which symptoms are exacerbated then have individuals perform supervised exercise at 80% of that rate,[3, 4] however this has not been done in the pediatric population and most pediatric physicians instead perform graduated activity protocols starting at a lower thresholds and increasing unless an exacerbation occurs (SORT Level of Evidence C).[5, 6] It is proposed that the fundamental cause of PCS is physiological dysfunction that fails to return to normal after a concussion. Essentially patients with a concussion are in a state of sympathetic nervous system predominance. This results in the subsequent altering of autonomic function and impaired cerebral auto regulation.[7] Aerobic exercise training may help concussion-related physiological dysfunction because exercise increases parasympathetic activity, reduces sympathetic activation, and improves cerebral blood flow. Recent articles have compared rest to activity and found slower recovery from PCS in most of the rest groups.[8]

The aim of this research is to provide documentation in the literature for an adolescent graduated activity protocol that is currently practiced in the University of Arizona Pediatric Sports Medicine Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 13 and 18 (freshman - senior)
2. Subject must be able to understand and sign assent form and parent/guardian must be able to understand and sign consent form
3. Initial injury meets the definition of mTBI as follows:

   a. Traumatically induced physiological disruption of brain function by at least one of the following: i. Any period of loss of consciousness of 30 minutes or less ii. Any loss of memory for events immediately before or after accident and post-traumatic amnesia not greater than 24 hours iii. Any alteration in mental state at time of accident b. No structural lesions in the head or brain
4. Diagnosed with post concussive syndrome as follows:

   a. Clinical SCAT-3 revised score of >22 at 3+ weeks or plateaued score for 2 weeks or more of >15 at 4+ weeks
5. Continues to experience symptoms post injury and at time of enrollment
6. Has had a normal MRI
7. Can commit to participating for 12 weeks

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from study participation:

1. Any documented structural lesions in the skull or brain
2. Borderline TBI or concern that TBI is moderate rather than mild
3. Any medication or condition that elevates heart rate

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in symptoms | 12 weeks
  Depression Anxiety Stress Scale and ImPACT Symptom Severity Scale

SECONDARY OUTCOMES:
Improvement in Neuropsychological testing performance | 12 Weeks
  ImPACT

CONTACTS AND LOCATIONS:
Overall Officials: Sydney A Rice, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Background] Harmon KG, Drezner JA, Gammons M, Guskiewicz KM, Halstead M, Herring SA, Kutcher JS, Pana A, Putukian M, Roberts WO. American Medical Society for Sports Medicine position statement: concussion in sport. Br J Sports Med. 2013 Jan;47(1):15-26. doi: 10.1136/bjsports-2012-091941. PMID 23243113
- [Background] Craton N, Leslie O. Is rest the best intervention for concussion? Lessons learned from the whiplash model. Curr Sports Med Rep. 2014 Jul-Aug;13(4):201-4. doi: 10.1249/JSR.0000000000000072. No abstract available. PMID 25014382
- [Background] Leddy JJ, Kozlowski K, Donnelly JP, Pendergast DR, Epstein LH, Willer B. A preliminary study of subsymptom threshold exercise training for refractory post-concussion syndrome. Clin J Sport Med. 2010 Jan;20(1):21-7. doi: 10.1097/JSM.0b013e3181c6c22c. PMID 20051730
- [Background] Schneider KJ, Iverson GL, Emery CA, McCrory P, Herring SA, Meeuwisse WH. The effects of rest and treatment following sport-related concussion: a systematic review of the literature. Br J Sports Med. 2013 Apr;47(5):304-7. doi: 10.1136/bjsports-2013-092190. PMID 23479489